CLINICAL TRIAL: NCT04535570
Title: Evolution of the Energy Expenditure During Hematopoietic Stem Cell Transplantation in Patients With Hematological Disease and Associated Factors
Brief Title: Evolution of the Energy Expenditure During Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Principal investigator, Federal University of Minas Gerais
Other Study IDs: 58010016.0.0000.5149
Record Dates: First submitted 2019-06-13; First posted 2020-09-02 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Bone Marrow Transplantation; Hematopoietic Stem Cell Transplantation
Keywords: Bone Marrow Transplantation; Hematopoietic Stem Cell Transplantation; Indirect Calorimetry; Energy Metabolism; Basal Metabolism
MeSH Terms: interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre Transplant: All 20 patients will have the energy expenditure measured in the pre-transplantation in order to compare with post-transplant data.
  Interventions: Other: Indirect Calorimetry
- Post Transplant: All 20 patients will have the energy expenditure measured in the post transplantation in order to compare with the pre-transplant data.
  Interventions: Other: Indirect Calorimetry

INTERVENTIONS:
Other: Indirect Calorimetry — In the pre-transplant, before the conditioning regime, and also on the 10th and 17th post-transplant, the resting energy expenditure was measured by indirect calorimetry.

SUMMARY:
The treatment before bone marrow transplantantion is initiated by chemotherapy associated or not with radiotherapy, both of which cause various side effects on the patient as symptoms that impair food intake. The nutritional status of the patient is one of the factors related to the success of the transplant, so a complete nutritional assessment before transplantation is necessary in order to identify patients at nutritional risk, nutritional disorders and to perform appropriate and early intervention to promote recovery and / or health maintenance. Will be used for nutritional assessment: arm perimeter, arm muscle area; electrical bioimpedance, phase angle, and Indirect Calorimetry, a standard method of noninvasive nutritional assessment that expresses the nutritional demand and rate of utilization of energy substrates from oxygen consumption and carbon dioxide production through the air inhaled and exhaled by the individual's lungs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological disease
* Age equal or superior to 15 years old
* Both sexes
* Will be submitted bone marrow transplantation

Exclusion Criteria:

* Age below 15 years old
* Those who can't perform calorimetry (oxygen therapy, mechanical ventilation)
* Have hyper or hypothyroidism
* Admitted to the Intensive Care Unit (without at least one result of post-transplant indirect calorimetry)
* Don't agree to participate in the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of both sexes, older than 15 years old, hospitalized in the Bone Marrow Transplant sector of the Hospital das Clínicas of the Federal University of Minas Gerais and submitted to transplantation will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | Up to 3 weeks after protocol termination
  The energy expenditure will be analyzed by the volume of oxygen (VO2) consumed, the volume of carbon dioxide (VCO2) produced and the respiratory quotient (VO2 / VCO2). The values analyzed will be the results of the measures of energy expenditure (BMR) before and after the transplant, in calories (Kcal), to verify changes caused by chemotherapy and / or radiation therapy.

SECONDARY OUTCOMES:
Nutritional status of patients | Up to 3 weeks after protocol termination
  We'll use ASG for this parameter. Patients will have nutritional status classified as malnourished, nourished or overweight, in the periods before and after transplantation to verify changes caused by chemotherapy and / or radiation therapy.
Caloric and protein adequacy | Up to 3 weeks after protocol termination
  The caloric and protein adequacy will be analyzed by the amount of calorie (kcal / kg / day) and protein (g / kg / day) intake, compared to calorie and protein required before and after transplantation, to verify changes caused by chemotherapy and / or radiation therapy.The caloric and protein adequacy will be presented with g/kg/day (protein) or kcal/kg/day (calories)
Clinical outcomes | Up to 3 weeks after protocol termination
  Patients will have the following outcomes:
  * constipation or diarrhea - Bristol stool scale pontuation (7 points scale)
  * mucositis (grade I-IV) - Dentistry report with grade of mucositis in grade I,II,III or IV
  * graft versus host disease (grade I-IV) - Medical report with grade of GVHD in grade I, II, III or IV
  * presence of Cytomegalovirus infection - Blood test Positive or Negative
  * colonization of Clostridium difficile - Feces Test Positive or Negative
  * infection by Candida - Laboratory test positive or negative
  * another diagnosis of infection - Medical report/ Yes or no for presence of this complication
  * presence of febrile neutropenia - Medical report / Yes or no for presence of this complication
  * length of hospital stay - number of complete days of hospitalization
  * death during the hospital stay - number of death during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Simone V Generoso, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Escola de Enfermagem - UFMG, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No